CLINICAL TRIAL: NCT02016248
Title: Prospective Evaluation of Stereotactic Body Radiotherapy Boost for Unfavorable Localized Prostate Cancer
Brief Title: SBRT Boost for Unfavorable Prostate Cancer'
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: MemorialCare Health System (Other)
Responsible Party: Principal Investigator, Asif Harsolia, MD, Radiation Oncologist, MemorialCare Health System
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 065-12
Record Dates: First submitted 2012-12-04; First posted 2013-12-19 (Estimated); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Prostate Cancer
Keywords: Boost; Prostate Cancer; Stereotactic Body Radiation; SBRT; Radiosurgery; SABR; Stereotactic Ablative Body Radiotherapy
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Radiosurgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment Arm (Experimental): All participants receive the same treatment: standard external-beam radiation therapy (EBRT) plus an SBRT boost.
  Interventions: Radiation: Stereotactic Body Radiotherapy

INTERVENTIONS:
Radiation: Stereotactic Body Radiotherapy — The intervention in this study is the SBRT boost, which is a short course of five high-dose stereotactic body radiotherapy treatments (5.5 Gy × 5 fractions, total 27.5 Gy) delivered with image-guided precision to the prostate. This SBRT boost is given in addition to standard external-beam radiation therapy (EBRT), which delivers 50.4 Gy to the pelvis, prostate, and proximal seminal vesicles.

SUMMARY:
The purpose of this study is to find out whether giving a short course of focused radiation called an SBRT "boost" is a safe and effective way to treat prostate cancer. This boost delivers a high dose of radiation to the prostate in a non-invasive way, similar to what is done with high dose rate (HDR) brachytherapy but without using needles. The study looks at how well this treatment controls the cancer, what side effects it may cause, and how it affects patients' quality of life over time.

DETAILED DESCRIPTION:
This study is designed to evaluate whether delivering a stereotactic body radiotherapy (SBRT) boost-a short course of five high-dose, precisely targeted radiation treatments-can safely and effectively replace the traditional invasive high dose rate (HDR) brachytherapy boost for men with unfavorable, high-risk, or very high-risk localized prostate cancer. The SBRT boost uses imaging-guided systems and gold fiducial markers to track prostate motion in real time, allowing submillimeter accuracy without placing needles inside the prostate. Treatment planning incorporates CT/MRI fusion, careful mapping of the urethra, and strict dose-volume limits for nearby organs such as the rectum and bladder to ensure the boost achieves HDR-equivalent tumor dosing while minimizing toxicity. All patients also receive standard external beam radiation therapy to the pelvis, and the combined course is designed based on biological dose modeling and prior HDR clinical experience to optimize tumor control while maintaining acceptable side-effect rates.

The protocol also includes structured follow-up and ongoing safety monitoring to track side effects, prostate-specific antigen (PSA) response, and quality-of-life outcomes. Patients are assessed at regular intervals-from two weeks post-treatment through five years-with physical exams, PSA testing, toxicity evaluations, and validated questionnaires measuring urinary and sexual function. Imaging such as prostate-specific membrane antigen (PSMA) PET/CT or bone scans is performed if biochemical failure or symptoms suggest disease progression. The study's primary goals are to determine the rate of significant gastrointestinal and genitourinary side effects and to measure biochemical disease-free survival at five years, while secondary goals include evaluating local and distant tumor control and longer-term survival outcomes. Stopping rules, adverse-event reporting procedures, and quality-assurance requirements are built into the protocol to ensure patient safety and regulatory compliance throughout the study.

ELIGIBILITY:
Inclusion

* Histologically proven prostate adenocarcinoma
* Biopsy within 12 months of date of registration required except for patients who already meet criteria for enrollment in the high risk arm of the protocol. For these patients, repeat biopsy will be at the discretion of the treating physician. In general, repeat biopsy is recommended for these patients, but is not required if it will not affect the treating physician's management decisions in regards to the care of the patient.
* Clinical Stage I-IV, MX-M0 (AJCC VERSION 9)
* M-stage determined by physical exam, CT, MRI, bone scan, PSMA PET/CT, or biopsy.
* Prostate volume: ≤ 100 cc (recommended not required)
* Determined using: volume = π/6 x length x height x width
* Measurement from CT, MRI or ultrasound ≤ 90 days prior to registration.
* Eastern Cooperative Oncology Group (ECOG) performance status 0-1
* No prior prostatectomy or cryotherapy of the prostate
* No prior radiotherapy to the prostate or lower pelvis
* No implanted hardware or other material that would prohibit appropriate treatment planning or treatment delivery, in the investigator's opinion.
* Completion of patient questionnaires in section 3.7.
* Consent signed

Exclusion

* No prior prostatectomy or cryotherapy of the prostate
* No prior radiotherapy to the prostate or lower pelvis
* No implanted hardware or other material that would prohibit appropriate treatment planning or treatment delivery, in the investigator's opinion.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2012-06 (Actual); Primary Completion 2028-06 (Estimated); Study Completion 2029-06 (Estimated)

PRIMARY OUTCOMES:
Rate of Grade 3-5 Gastrointestinal (GI) and Genitourinary (GU) Toxicities | 5 years
  This outcome measures how many participants experience severe (grade 3-5) side effects involving the gastrointestinal or genitourinary systems after receiving the SBRT boost. Toxicities are evaluated using the NCI Common Terminology Criteria for Adverse Events (CTCAE).

SECONDARY OUTCOMES:
Local Failure Rate | 10 years
  The study looks at whether the cancer comes back in the prostate or spreads elsewhere, how long patients stay cancer-free, and how long they live with or without prostate cancer. It also measures overall survival from any cause and tracks changes in urinary and sexual function using brief questionnaires over time. These outcomes are monitored throughout regular follow-up visits for up to 5 years, with some patients followed as long as 10 years if the investigators choose to continue long-term monitoring.

CONTACTS AND LOCATIONS:
Overall Officials: Asif Harsolia, MD, Principal Investigator — MemorialCare
Locations (3):
- United States (3):
  - Orange Coast Memorial Medical Center, Fountain Valley, California
  - Saddleback Memorial Medical Center, Laguna Hills, California
  - Long Beach Memorial Medical Center, Long Beach, California